CLINICAL TRIAL: NCT03491163
Title: Evaluation of Damaging Factors to Endothelial Glycocalyx During On-pump Coronary Artery Bypass Surgery
Brief Title: Evaluation of Damaging Factors to Endothelial Glycocalyx During Heart Surgery Pilot Study
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Tadas Cesnaitis (Other)
Responsible Party: Sponsor-Investigator, Tadas Cesnaitis, PhD student, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Other Study IDs: ENDOTEL SYNDECAN-1
Record Dates: First submitted 2018-03-29; First posted 2018-04-09 (Actual); Last update posted 2018-08-07 (Actual); Status verified 2018-08

CONDITIONS: Heart; Surgery, Heart, Functional Disturbance as Result
Keywords: syndecan-1; endothelial glycocalyx; On-pump heart surgery

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients: Syndecan-1 concentration evaluation
  Interventions: Diagnostic Test: Syndecan-1 concentration evaluation

INTERVENTIONS:
Diagnostic Test: Syndecan-1 concentration evaluation — Blood sample will be taken and analysed using ELISA method.

SUMMARY:
Evaluation of endothelial glycocalyx damage in on-pump conventional coronary artery bypass surgery using a syndecan-1 (CD138) blood test. The study will be carried out in two stages. Pilot study for testing and correcting research methodology and the main study.

DETAILED DESCRIPTION:
Study tasks:

1. To evaluate changes of syndecan-1 concentration during surgery and postoperative period.
2. Determine the effect of aortic clamping and on-pump duration on endothelial glycocalyx damage.
3. Assess the risk of early postoperative complications and syndecan-1 plasma concentrations.
4. To evaluate the correlation of inflammatory status with glycocalyx damage.
5. To evaluate glycocalyx damage to patients with diabetes vs non-diabetes.

Methods:

Patients undergoing cardiopulmonary bypass surgery are being treated at the Heart, Chest and Vascular Surgery Clinic of the Lithuanian University of Health Sciences Hospital in Kaunas Clinics. After receiving patients written consent a syndecan-1 concentration test will be performed upon arrival at the operating room, before cardiopulmonary bypass (CPB), after CPB, upon arrival in the ICU and after 24 hours.

All needed data for evaluating patients outcome will be taken from medical documentation during patients stay in hospital.

ELIGIBILITY:
Inclusion Criteria:

* Elective on-pump coronary artery bypass surgery needed.
* Normal heart function at the time of operation.
* Patients without infections.
* Patients who signed study informed consent form

Exclusion Criteria:

* Life saving operation.
* Renal or hepatic dysfunction.
* Off-pump heart operation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: People with normal or compensated heart function, with normal inflammatory status, who have agreed to participate in the study. Patients undergoing elective on-pump coronary artery bypass surgery.
Sampling Method: Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2018-03-29 (Actual); Primary Completion 2019-10-30 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
Changes of syndecan-1 concentration during surgery and postoperative period. | 2 years
  Concentration of syndecan-1 will be measured by taking patients blood sample before operation, after aortic cannulation, after CPB, when arriving to ICU and 24 hours after operation. Means of concentration changes will be compared to determine which period of operation has the biggest impact to endothelial glycocalyx shedding.
The evaluation of aortic clamping and on-pump duration on endothelial glycocalyx damage using syndecan-1 concentration measure. | 2 years
  Concentrations of syndecan-1 will be evaluated considering the duration of aortic clamping and CPB. Optimal duration will be searched for minimal impact to endothelial glycocalyx.
Assess the risk of early postoperative complications and find possible correlation to syndecan-1 concentration changes. | 2 years
  All negative events after operation will be recorded and statistically correlated with syndecan-1 concentration changes.
The correlation of inflammatory status with glycocalyx damage. | 2 years
  Leucocytosis and C reactive protein levels will be evaluated before, after heart operation and 24 hours later. Data will be compared to syndecan-1 concentration changes.
Glycocalyx damage to patients with diabetes vs non-diabetes during heart surgery. | 2 years
  Compare glycocalyx damage using syndecan-1 concentration changes to diabetic and non-diabetic patents during heart surgery.

CONTACTS AND LOCATIONS:
Overall Officials: Edmundas Sirvinskas, Prof, Principal Investigator — Professor at Lithuanian University of Health Sciences
Locations (1):
- Lithuanian University of Health Sciences, Kaunas, Lithuania

IPD SHARING:
Plan to Share IPD: No